CLINICAL TRIAL: NCT07161544
Title: An Open-label, Multicenter, Two Part, Ascending Dose Followed by a Controlled Trial to Assess the Safety and Efficacy of a Subretinal Administration of AAVB-039 in Participants With Stargardt Disease (STGD1) (CELESTE)
Brief Title: A Study of AAVB-039 in Participants With Stargardt Disease (STGD1)
Acronym: CELESTE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AAVantgarde Bio Srl (Industry)
Collaborators: AAVantgarde Bio UK Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 039-101
Record Dates: First submitted 2025-08-08; First posted 2025-09-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Stargardt Disease
Keywords: Stargardt Disease; Biallelic Mutation; Gene Mutation; ABCA4
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): AAVB-039 dose level 1 (low dose)
  Interventions: Biological: AAVB-039
- Cohort 2 (Experimental): AAVB-039 dose level 2 (mid dose)
  Interventions: Biological: AAVB-039
- Cohort 3 (Experimental): AAVB-039 dose level 3 (high dose)
  Interventions: Biological: AAVB-039
- Cohorts 4-5 (Experimental): AAVB-039 dose level 1, 2 or 3
  Interventions: Biological: AAVB-039

INTERVENTIONS:
Biological: AAVB-039 — Single subretinal administration

SUMMARY:
The purpose of the 039-101 study is to evaluate the safety and tolerability of a single subretinal injection of AAVB-039 in participants with Stargardt disease secondary to a biallelic mutation of the ABCA4 gene. The study will also assess initial efficacy following AAVB-039 administration.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of Stargardt disease due to ABCA4 mutation
* Willingness to adhere to protocol per informed consent

Exclusion Criteria:

* Unwillingness to meet the requirements of the study
* Participation in a clinical study with another Investigation Medicinal Product
* Previous participation in another gene or cell therapy trial
* Any condition that would preclude subretinal surgery
* Complicating ocular and/or systemic diseases

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2032-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
To measure the number and severity of treatment related adverse events following treatment with AAVB-039 | 0-60 months

SECONDARY OUTCOMES:
Change in the area of atrophy (assessed via short wavelength fundus autofluorescence (SW-FAF), following treatment with AAVB-039 | 0-60 months
Change in ellipsoid zone (EZ) loss following treatment with AAVB-039 | 0-60 months
Change in macular sensitivity assessed via microperimetry following treatment with AAVB-039 | 0-60 months
Change in visual acuity following treatment with AAVB-039 | 0-60 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
- United Kingdom (2):
  - Moorfields Eye Hospital NHS Foundation Trust, London, England
  - The Retina Clinic, London, England

IPD SHARING:
Plan to Share IPD: No